CLINICAL TRIAL: NCT05883813
Title: Immediate Effects of Suboccipital Muscle Release Combined With Sustained Natural Apophyseal Glides in Patients With Chronic Tension Type Headache
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Foundation University Islamabad (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FUI/CTR/2023/11
Record Dates: First submitted 2023-05-22; First posted 2023-06-01 (Actual); Last update posted 2023-06-01 (Actual); Status verified 2023-05

CONDITIONS: Tension-Type Headache
MeSH Terms: conditions — Tension-Type Headache

STUDY DESIGN:
Intervention Model Description: This study is randomized controlled trial which consist of 2 groups. One group will be given suboccipital muscle release. Second group will be given SNAGS along with sub-occipital muscle release. All the groups were recruited concurrently.
Who Masked: Participant
Masking Description: The participant does not know about the group in which he is included.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Active Comparator): suboccipital muscle release for 10 mins + 5 min general warm up exercises + 10 min hot pack + 10 min TENS + trapezius stretching with 3 sec hold and 5 reps
  Interventions: Procedure: suboccipital muscle release; Procedure: Supplemental therapy
- Group 2 (Experimental): suboccipital muscle release for 10 mins + SNAGS: 3 glides with 10 sec hold of each glide + 5 min general warm up exercises + 10 min hot pack + 10 min TENS + trapezius stretching with 10 sec hold and 5 reps
  Interventions: Procedure: sustained natural apophyseal glides (SNAGS); Procedure: suboccipital muscle release; Procedure: Supplemental therapy

INTERVENTIONS:
Procedure: sustained natural apophyseal glides (SNAGS) — SNAGS will be given with patient in sitting position and the therapist will be standing behind the patient. The therapist will place the thumb on the spinous process of the vertebra. Move spinous process upward towards the eyeball direction & maintain the glide and ask the patient to turn (rotation) his head slowly in painful direction, sustain the mobilization until head turn to the midline. Three repetitions of each glide will be given and each glide will be maintained for 10 seconds at end range.
  Arms: Group 2
Procedure: suboccipital muscle release — Sub-occipital muscle release will be applied with the patient in the supine position with the eyes closed and the physiotherapist's hands placed under the patient's head, in contact with the sub-occipital muscles. The physiotherapist progressively increased the pressure exerted during the 10 minutes of treatment.
Procedure: Supplemental therapy — General warm-up exercises, TENS, hot pack, trapezius stretching

SUMMARY:
Headache disorder characterized by recurrent headache are among the most common disoredrs of the nervous system. Tension type headache is widely recognized kind of headache that affects 80% of the individuals. Its underlying cause has not been clearly distinguished. It is managed both pharmacology and non-pharmacology which includes dry needling, acupuncture, manual techniques and massage. Several studies conducted which showed that both the soft tissue muscle inhibition and joint mobilization techniques are effective in decreasing pain. But there is lack of evidence which shows combined effects of soft tissue muscle inhibition and sustained natural apophyseal glides(SNAGS) in chronic tension type headache. so this study will compare the effects of soft tissue muscle release and SNAGS on pain intensity and cervical range of motion.

DETAILED DESCRIPTION:
Headache disorder characterized by recurrent headache are among the most common disoredrs of the nervous system. Tension type headache is one of the widely recognized kind of headache that affects 80% of the individuals. Its underlying cause has not been clearly distinguished.Chronic tension type headache causes tightness in the suboccipital muscle which may result in decrese in range of motion in cervical region. It is managed both pharmacology and non-pharmacology which includes dry needling, acupuncture, manual techniques and massage. Several studies conducted which showed that both the soft tissue muscle inhibition and joint mobilization techniques are effective in decreasing pain. But there is lack of evidence which shows combined effects of soft tissue muscle inhibition and sustained natural apophyseal glides(SNAGS) in chronic tension type headache. so this study will compare the effects of soft tissue muscle release and SNAGS on pain intensity and cervical range of motion.

This study will be conducted in fauji foundation hospital using non-probability purposive sampling technique. Sample size calaculated from open epi tool is 48, with 24 patients in each group. Patients are selected on the basis of inclusion criteria. Patients will be guided about the benefits and risks of the study, right to withdraw from the study at any point and confidentiality of the data. After diagnosis by the physician according to the ICHD-3 criteria, written consent will be taken from each participant. Then they randomly assigned into 2 groups via lottery method. Cervical range of motion, blood pressure and pain intensity will be measured before and after the treatment. Suboccipital muscle release and SNAGS will be given to experimental group and suboccipital muscle release only to the control group.

Group 1(Control group): suboccipital muscle release for 10 mins + 5 min general warm up exercises + 10 min hot pack + 10 min TENS + trapezius stretching with 3 sec hold and 5 reps.

Group 2(Experimental group): suboccipital muscle release for 10 mins + SNAGS: 3 glides with 10 sec hold of each glide + 5 min general warm up exercises + 10 min hot pack + 10 min TENS + trapezius stretching with 10 sec hold and 5 reps.

Sub-occipital muscle release: This technique will be performed in the supine position with the patient's eyes closed and the physiotherapist's hands placed under the patient's head, in contact with the sub-occipital muscles. The physiotherapist progressively increased the pressure exerted during the 10 minutes of treatment.

SNAGS: This technique will be performed with patient in sitting position and the therapist may be standing behind the patient. The therapist would place the thumb on the spinous process of the vertebra. Move spinous process upward towards the eyeball direction & maintain the glide and ask the patient to turn (rotation) his head slowly in painful direction, sustain the mobilization until head turn to the midline. Three repetitions of each glide were given and maintain for 10 seconds at end range.

Pain intensity, cervical range of motion and blood pressure will be measured immediately after the treatment.

ELIGIBILITY:
Inclusion Criteria:

* 18-64 years old
* Male and Female
* International classification of headache disorders-3 diagnosis:
* Headache occurring on 15 days/month on average for >3 months (180 days/year),
* Lasting hours to days, or unremitting -At least two of the following four characteristics:-
* Bilateral location
* Pressing or tightening (non-pulsating) quality
* Mild or moderate intensity
* Not aggravated by routine physical activity such as walking or climbing stairs
* Both of the following:
* No more than one of photophobia, phonophobia or mild nausea
* Neither moderate or severe nausea nor vomiting
* Not better accounted for by another ICHD-3 diagnosis.

Exclusion Criteria:

* Patients with other types of primary or secondary headache e.g cervicogenic headache
* History of trauma to the cervical spine
* Vertigo, dizziness, uncompensated neck tension
* Spurling test positive
* Flexion compression test positive
* Extension compression test positive
* Cervical flexion rotation test positive
* Pregnancy

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-06-15 (Estimated); Study Completion 2023-07-01 (Estimated)

PRIMARY OUTCOMES:
cervical range of motion | Immediate after treatment
  The cervical range of motion will be measured by using goniometer. The patient will be in sitting position. For flexion and extension, the fulcrum will be placed on external auditory meatus, the stationary arm will be vertical to the ground with moving arm aligned parallel with the base of the ear. For side bending, the fulcrum will be placed on C7 vertebrae, the stationary arm perpendicular to the ground and moving arm parallel to the external occipital protuberence. For rotation, the fulcrum will be placed on the central cranial aspect of head, stationary arm parallel to the acromion process and moving arm align with tip of the nose. The angle between the stationary and moving arm will be measured.

SECONDARY OUTCOMES:
Pain intensity | Immediate after treatment
  Will be measured with NPRS
Blood pressure | Immediate after treatment
  Will be measured with sphygmomanometer

CONTACTS AND LOCATIONS:
Locations (1):
- Fauji Foundation Hospital, Rawalpindi, Punjab Province, Pakistan